CLINICAL TRIAL: NCT05061264
Title: Complex Abdominal Wall Reconstruction With Polyvinylidene (PVDF) Mesh in the Setting of Active Infection: a Prospective Case-control Series.
Brief Title: Abdominal Wall Reconstruction With PVDF Mesh in the Setting of Active Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Claudio Birolini, MD, phD. Director of General Surgery of the Third Division of Clinical Surgery of the Department of Surgery, Head of the Hernias and Abdominal Wall Group, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVDF mesh
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Wall Defect; Abdominal Wall Hernia; Abdominal Wall Infection; Abdominal Wall Fistula; Infection
Keywords: ventral hernia; mesh infection; enteric fistula; polyvinylidene mesh; synthetic mesh; abdominal wall reconstruction; complex hernia; DynaMesh
MeSH Terms: conditions — Hernia, Abdominal; Infections; Hernia, Ventral | interventions — Abdominoplasty

STUDY DESIGN:
Intervention Model Description: A study group submitted to abdominal wall repair with PVDF mesh in the infected setting compared to a control group submitted to abdominal wall repair with PVDF mesh in the clean setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active infection group (Experimental): A cohort of 38 patients carrying an active infection (mesh sinus, exposed mesh or enteric fistulas) resulting from a previous hernia repair, with or without an associated recurrent ventral hernia, and submitted to abdominal wall reconstruction with PVDF mesh.
  Interventions: Procedure: Abdominal wall reconstruction
- Clean control group (Active Comparator): A cohort of 38 patients with ventral hernias, and submitted to clean ventral hernia repair with PVDF mesh.
  Interventions: Procedure: Abdominal wall reconstruction

INTERVENTIONS:
Procedure: Abdominal wall reconstruction — The repair of abdominal wall defects with polyvinylidene (PVDF) mesh
  Other Names: Ventral hernia repair

SUMMARY:
The use of synthetic mesh to repair infected defects of the abdominal wall remains controversial. This study aimed to evaluate the short-term outcomes of using PVDF mesh to treat infected abdominal wall defects in the elective setting.

DETAILED DESCRIPTION:
From May 2016 until February 2021, 38 patients presenting with chronic mesh infection and/or enteric fistulas were enrolled in this prospective study. The active infection group (AI) was compared to a cohort of 38 patients submitted to clean ventral hernia repairs (CC). The inclusion criteria in the AI group were the presence of active chronic mesh infection (non-healing sinus, exposed mesh, or mesh-related enteric fistulas) resulting from a previous repair, or the presence of an enteric/enteroatmospheric fistula, with or without an associated abdominal wall defect. The patients invited to participate as controls had a primary or recurrent ventral hernia without previous history of infection and were eligible for clean operations. The operations in the AI group were classified as Class IV (dirty-infected), according to the CDC Wound Classifications, as adopted by the European registry for abdominal wall hernias.

The exclusion criteria were giant ventral hernias, patients on immunosuppressive or corticosteroid therapy, patients with portal hypertension, Crohn's disease, acute postoperative mesh infection, chronic infections following inguinal hernia repair, and emergency operations.

Demographic data included age, gender, American Society of Anesthesiologists (ASA) score, body mass index (BMI), comorbidities, smoking status, cancer history, and the number of previous abdominal operations. Perioperative details included the list of associated procedures, the defect width, the extension of the pre-aponeurotic dissection, operative time, and anesthesia time. Further analysis in the AI group included the clinical presentation, the onset of symptoms, the type and position of the infected mesh, the possible causes for mesh infection, and the microbiology of mesh explants.

Patients were followed and operated at the Abdominal Wall and Hernia Repair Unit at the Hospital das Clínicas, University of São Paulo, Brazil. Six surgeons of the team conducted the operations in both groups. The local ethics committee approved the study. Informed consent was obtained from all individual participants. The study was registered at the national registry, Plataforma Brasil (https://plataformabrasil.saude.gov.br/login.jsf), CAAE 52383615.0.0000.0068, and Identifier 1.412.367.

All the mesh samples used were provided by the manufacturer (FEG Textiltechnik, Aachen, Germany) through their local dealer (BMR Medical, www.bmrmedical.com.br), at no cost. None of the authors or our institution received any financial support to undertake the study.

The primary outcomes were the presence of any surgical site occurrences (SSO) or surgical site infection (SSI) during the first 30 days after the operation. The secondary outcomes included developing hernia recurrence or the recurrence of mesh infection during a 6-month follow-up period. An SSI was defined as an infection occurring where the surgery took place and was further defined as superficial, deep, and organ space. An SSO was described as any surgical infection, wound breakdown, soft tissue ischemia, seroma, and hematoma formation. A surgical site occurrence requiring procedural intervention (SSOPI) was described as any wound event requiring the opening of the wound, wound debridement, suture excision, percutaneous drainage, hematoma evacuation, or mesh removal [14]. The Clavien-Dindo classification [15] (Table 2) was applied to all surgical complications. Suspected recurrences of a hernia or infection were determined by physical examination and CT scan imaging. Non-surgical complications, other operations, and deaths were recorded during the follow-up period.

The statistical analysis was performed using the computer software Stata: version 16.0 (Stata Corp. 2019. Stata: Release 16. Statistical Software. College Station, TX: Stata Corp LLC). The frequency distribution was used by means to describe categorical variables (number of cases and relative percentage) and for continuous variables, measures of central tendency (median and mean) and variability (range and standard deviation). The nonparametric Mann-Whitney U test was applied for the statistical evaluation of the association between groups and continuous variables. The Student t-test was adopted when data normality was identified. Shapiro-Wilk test was applied to verify the normality of data. The association between categorical variables in contingency tables was analyzed using the frequency Chi-square test and the Fisher exact test adopted in 2x2 tables whenever at least one expected frequency was less than five. The 5% significance level was considered for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Study group: patients with the presence of an active chronic mesh infection (non-healing sinus, exposed mesh, or mesh-related enteric fistulas) resulting from a previous repair, or the presence of an enteric/enteroatmospheric fistula, with or without an associated abdominal wall defect
* Control group: patients with a primary or recurrent ventral hernia without previous history of infection and eligible for clean operations

Exclusion Criteria:

* giant ventral hernias with a volume ratio higher than 25% and loss of domicile
* patients on immunosuppressive therapy or using corticosteroids
* patients with portal hypertension
* patients with Chron´s disease
* acute postoperative mesh infection
* chronic mesh infections following inguinal hernia repair
* emergency operations.

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Surgical site occurence | 30 days
  any surgical infection, wound breakdown, soft tissue ischemia, seroma, and hematoma formation
Surgical site infection | 30 days
  as an infection occurring where the surgery took place and was further defined as superficial, deep, and organ space

SECONDARY OUTCOMES:
Hernia recurrence | 6 and 36 months
  the recurrence of an incisional hernia
Infection recurrence | 6 and 36 months
  the recurrence of a chronic infection, or mesh related infection

OTHER OUTCOMES:
Microbiology of mesh infection | 30 days
  the study of the microorganisms causing chronic infection

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Birolini, MD, Principal Investigator — Hospital das Clinicas da FMUSP
Locations (1):
- Hospital das Clinicas da FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Patient records and pictures, both of the operations and follow up data, are available.
Supporting Information: CSR
Time Frame: From september 2021, available for 1 year
Access Criteria: Available data to be shared with researchers interested in abdominal wall reconstruction

REFERENCES:
- [Background] Birolini C, de Miranda JS, Tanaka EY, Utiyama EM, Rasslan S, Birolini D. The use of synthetic mesh in contaminated and infected abdominal wall repairs: challenging the dogma-A long-term prospective clinical trial. Hernia. 2020 Apr;24(2):307-323. doi: 10.1007/s10029-019-02035-2. Epub 2019 Sep 6. PMID 31493051
- [Background] Klinge U, Klosterhalfen B, Ottinger AP, Junge K, Schumpelick V. PVDF as a new polymer for the construction of surgical meshes. Biomaterials. 2002 Aug;23(16):3487-93. doi: 10.1016/s0142-9612(02)00070-4. PMID 12099293
- [Background] Garner JS. CDC guideline for prevention of surgical wound infections, 1985. Supersedes guideline for prevention of surgical wound infections published in 1982. (Originally published in November 1985). Revised. Infect Control. 1986 Mar;7(3):193-200. doi: 10.1017/s0195941700064080. No abstract available. PMID 3633903
- [Background] Haskins IN, Horne CM, Krpata DM, Prabhu AS, Tastaldi L, Perez AJ, Rosenblatt S, Poulose BK, Rosen MJ. A call for standardization of wound events reporting following ventral hernia repair. Hernia. 2018 Oct;22(5):729-736. doi: 10.1007/s10029-018-1748-6. Epub 2018 Feb 10. PMID 29429064
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Hodgkinson JD, Maeda Y, Leo CA, Warusavitarne J, Vaizey CJ. Complex abdominal wall reconstruction in the setting of active infection and contamination: a systematic review of hernia and fistula recurrence rates. Colorectal Dis. 2017 Apr;19(4):319-330. doi: 10.1111/codi.13609. PMID 28102927
- [Derived] Birolini C, Faro Junior MP, Terhoch CB, de Miranda JS, Tanaka EY, Utiyama EM. Microbiology of chronic mesh infection. Hernia. 2023 Aug;27(4):1017-1023. doi: 10.1007/s10029-023-02747-6. Epub 2023 Feb 9. PMID 36757611